CLINICAL TRIAL: NCT02263599
Title: Conservative Treatment For Ventral Hernia
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Frederik Helgstrand, MD, Zealand University Hospital
Other Study IDs: DK_01
Record Dates: First submitted 2014-09-20; First posted 2014-10-13 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Conservatively treated ventral hernias
- Surgically treated ventral hernias

SUMMARY:
The aim of this study is to evaluate on which indication patients are offered operative treatment for their ventral hernia, and to investigate the natural course of ventral hernia in the population of patients not offered operation.

ELIGIBILITY:
Inclusion Criteria:

All patients (older than 18 years) referred to the Surgical Department of Køge University Hospital from 2009 - 2014 with the diagnosis ventral hernia

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to the Surgical Department of Køge University Hospital in the timeperiod from 2009 - 2014 with the diagnosis ventral hernia
Sampling Method: Non-Probability Sample
Enrollment: 2089 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percentage of conservatively treated ventral hernias that undergo surgery | 5 years
  Percentage of conservatively treated ventral hernias at the primary surgical consultation, that undergoes surgery (acute or elective) later on

SECONDARY OUTCOMES:
Percentage of patient with ventral hernia that are treated conservatively | 5 years
  Percentage of patient referred to Køge Surgical Department with ventral hernia that are treated conservatively instead of surgically

CONTACTS AND LOCATIONS:
Overall Officials: Dunja Kokotovic, MS, Principal Investigator — Dept. of Surgery, Køge Hospital
Locations (1):
- Dept. of Surgery, Køge University Hospital, Køge, Denmark